CLINICAL TRIAL: NCT01380431
Title: Randomized, Open-label, Three Treatment Crossover Comparative Bioavailability Study of Lisinopril Tablets, 40 mg - Effect of Food Study
Brief Title: A Comparative Bioavailability Study of Lisinopril Tablets, 40 mg - Effect of Food Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: PharmaKinetics Laboratories Inc. (Industry)
Responsible Party: Alfred Elvin/Director of Biopharmaceutics, Par Pharmaceutical, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 11508
Record Dates: First submitted 2008-04-01; First posted 2011-06-27 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: To Determine Bioequivalence Under Fed Conditions
Keywords: bioequivalence, lisinopril, fed
MeSH Terms: conditions — Lecithin Cholesterol Acyltransferase Deficiency | interventions — Lisinopril; Tablets; Single Person

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Subjects received the Par formulated product.
  Interventions: Drug: Lisinopril
- B (Active Comparator): Subjects received the IPR (Zeneca Pharmaceuticals) formulated product.
  Interventions: Drug: lisinopril
- C (Active Comparator): Subjects received the IPR (Zeneca Pharmaceuticals) formulated product.
  Interventions: Drug: Lisinopril

INTERVENTIONS:
Drug: Lisinopril — Tablets, 40 mg, single oral dose
  Other Names: Zestril (R) Tablets, 40 mg, single, oral dose
  Arms: C
Drug: lisinopril — Tablets, 40 mg, single, oral dose
  Other Names: Zestril (R) Tablets, 40 mg, single, oral dose
  Arms: B
Drug: Lisinopril — 50% of subjects received the Par formulated product.
  Other Names: Zestril (R) Tablets, 40 mg, single, oral dose
  Arms: A

SUMMARY:
The purpose of this study is to compare the bioavailability of Par Lisinopril 40 mg Tablets and IPR Pharmaceuticals, Inc. Zestril (R).

DETAILED DESCRIPTION:
To compare the bioavailability of Par Lisinopril 40 mg Tablets and IPR Pharmaceuticals, Inc. Zestril (R), 40 mg - Effect of Food Study

ELIGIBILITY:
Inclusion Criteria:

* Males, healthy, 18-50 years of age,
* No more than plus or minus 15% from ideal weight for subject's height as defined by Metropolitan Life Insurance Company Statistical Bulletin 1983,
* Without a history of asthma, angioedema, hypertension, psychiatric illness, organ-system (cardiovascular, neurological, hematopoietic, renal, pulmonary, endocrine, or gastrointestinal,) disorders, ongoing infectious diseases, alcohol or drug abuse as determined by a medical history and/or physical examination within 30 days prior to the start of the study. Deviations may be acceptable if deemed not clinically significant by the investigator.
* Blood chemistry (including alkaline phosphatase, glucose, ALt, AST, LDH, BUN, GGT, creatinine, bilirubin, electrolytes), hematology (including hemoglobin, hematocrit, red blood cell count, white blood cell count, differential, platelet count), and urinalysis values within clinically acceptable limits upon evaluation by the investigator. The above tests will be performed within 30 days prior to the start of the study.
* No prescription drugs within 14 days, or OTC preparations (with the exception of acetaminophen, vitamins, medicated lozenges, dietary supplements and topical medications) within 7 days of the first drug administration, each period. Deviations may be acceptable if evaluated by the investigator and determined not to be clinically significant.
* No alcohol consumption for at least 48 hours prior to drug administration until after the last blood collection, each period.
* No known allergy to lisinopril or other ACE (angiotensin converting enzyme) inhibitors, such as captopril and enalapril, or to atropine.
* Acceptable electrocardiogram: sinus rhythm with no evidence of AV block or ischemic changes.
* At screening and check-in for each period, subjects must have blood pressure and pulse rate within the following ranges: Systolic blood pressure (110-150 mmHg); Diastolic blood pressure (70-95 mmHg); Pulse (50-105 bpm). Minor deviations (1-3 mmHg) at check-in may be acceptable at the discretion of the physician investigator. For all except the first period check-in, if a subject's vital signs measurements fall outside the range specified above, the subject may, at the discretion of the physician investigator, be allowed to remain enrolled until 0-hour measurements are made. If the 0-hour protocol vital signs requirements are met, the investigator may allow dosing and the subject's continuation in the study. If 0-hour vital signs requirements are not met, the subject will not be dosed and must be withdrawn from the study. The blood pressure and pulse will be measured after the subject has been seated at least three minutes. Subjects with blood pressure and pulse measurements outside the ranges will have their vital signs measurements repeated according to Standard Operating Procedure.
* No caffeine for at least 48 hours prior to dosing until after the last blood collection, each period.
* Negative HIV 1, hepatitis B surface antigen and urine screen for drugs of abuse within 30 days prior to the start of the study.

Exclusion Criteria:

* All Females, and males younger than 18 years of age or older than 50 years of age are not eligible to participate in this study.
* A weight that is more than plus or minus 15% from ideal weight for subject's height as defined by Metropolitan Life Insurance Company Statistical Bulletin 1983.
* A medical history of asthma, angioedema hypertension, psychiatric illness, organ-system (cardiovascular, neurological, hepatic, hematopoietic, renal, pulmonary, endocrine, or gastrointestinal) disorders, ongoing infectious diseases, alcohol or drug abuse within 30 days prior to start of the study.
* Blood chemistry (including alkaline phosphatase, glucose, ALt, AST, LDH, BUN, GGT, creatinine, bilirubin, electrolytes), hematology (including hemoglobin, hematocrit, red blood cell count, white blood cell count, differential, platelet count), and urinalysis values not within clinically acceptable limits upon evaluation by the investigator. The above tests will be performed within 30 days prior to the start of the study.
* Evidence of usage of prescription drugs within 14 days, or OTC preparations (with the exception of acetaminophen, vitamins, medicated lozenges, dietary supplements and topical medications) within 7 days of the first drug administration, each period.
* Alcohol consumption within 48 hours prior to drug administration until.
* Known allergy to lisinopril or other ACE (angiotensin converting enzyme) inhibitors, such as captopril and enalapril, or to atropine.
* Unacceptable electrocardiogram: sinus rhythm with evidence of AV block or ischemic changes.
* Blood pressure and pulse rate outside of the following ranges: Systolic blood pressure (110-150 mmHg); Diastolic blood pressure (70-95 mmHg); Pulse (50-105 bpm).
* Evidence of caffeine use within the last 48 hours, prior to dosing, or through the study up to and after the last blood collection, each period.
* A positive HIV 1, hepatitis B surface antigen and urine screen for drugs of abuse within 30 days prior to the start of the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 1999-08; Primary Completion 1999-10 (Actual); Study Completion 1999-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence
  Comparable food effect; The ratios of the test nd reference means and geometric means using the lease-squares means AUCo-t, AUCo-inf and Cmax should be within 80% - 125%.

CONTACTS AND LOCATIONS:
Overall Officials: Clifford L Ferguson, MD, Principal Investigator — PharmaKinetics Laboratories Inc.
Locations (1):
- PharmaKinetics Laboratories, Inc., Baltimore, Maryland, United States